CLINICAL TRIAL: NCT04180735
Title: Intestinal Perforation in Patients Receiving an Orthtopic Liver Transplantation in the Montpellier University Hospital: a Retrospective and Observational Study.
Brief Title: Intestinal Perforation in Patients Receiving an Orthtopic Liver Transplantation in the Montpellier University Hospital
Acronym: Perfogreffe
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Université Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0362
Record Dates: First submitted 2019-08-06; First posted 2019-11-29 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-08

CONDITIONS: Liver Transplantation; Intestinal Perforation; Digestive System Fistula; Intestinal Fistula
Keywords: Risk Factors; Survival
MeSH Terms: conditions — Intestinal Perforation; Digestive System Fistula; Intestinal Fistula | interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Perforation: Perforation
  Interventions: Procedure: Liver transplantation
- No perforation: No perforation
  Interventions: Procedure: Liver transplantation

INTERVENTIONS:
Procedure: Liver transplantation — Liver transplantation

SUMMARY:
Liver transplantation enhances the prognosis of patients with cirrhoses or hepatocellular carcinoma. However some patients develop intestinal perforations for which the prognosis is poor.

The aim of the study is to evaluate the risk factors of intestinal perforations using a retrospective study scheme.

DETAILED DESCRIPTION:
Liver transplantation enhances the prognosis of patients with cirrhoses or hepatocellular carcinoma. However some patients develop intestinal perforations for which the prognosis is poor.

The aim of the study is to evaluate the risk factors of intestinal perforations using a retrospective study scheme. Previous studies have shown a possible implication of drugs or medical history or intraoperative complications. The investigators aim to describe the other possible risk factors (such as portal vein clampage) and the type of surgery done after the diagnosis and its impact on survival as well.

ELIGIBILITY:
Inclusion Criteria:

* Patients having received an orthotopic liver transplantation in the Montpellier University Hospital from 2014 to 2019
* for the group Perforation: patients having during the follow-up a complication such as intestinal perforation. The complete list uses the ICD-10 codes for intestinal perforation, esophageal perforation, duodenal perforation etc.

Exclusion Criteria:

* No exclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having received an orthotopic liver transplantation in the Montpellier University Hospital from 2014 to 2019
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the total length of stay | 1 month
  Evaluate the total length of stay
Evaluate the total length of stay | 3 months
  Evaluate the total length of stay
Evaluate the total length of stay | 6 months.
  Evaluate the total length of stay

SECONDARY OUTCOMES:
Evaluate the occurrence of death | 1 month, 3 months, 6 months.
  Evaluate the occurrence of death
Evaluate the total number of complications | 1 month, 3 months, 6 months.
  Evaluate the total number of complications
Evaluate the number of perforations | 1 month, 3 months, 6 months.
  Evaluate the number of perforations
Evaluate the quality of life | 1 month, 3 months, 6 months.
  Evaluate the quality of life
Evaluate the occurrence of an acute or chronic rejection | 1 month, 3 months, 6 months.
  Evaluate the occurrence of an acute or chronic rejection

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio PANARO, PhD, Study Director — UH MONTPELLIER
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC